CLINICAL TRIAL: NCT00002158
Title: Open-Label Compassionate Use of Nitazoxanide for the Treatment of Cryptosporidiosis in AIDS Patients
Brief Title: A Study to Evaluate the Use of Nitazoxanide to Treat Cryptosporidiosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Romark Laboratories L.C. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 253B; UMD-95-009
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: Cryptosporidiosis; Diarrhea; Acquired Immunodeficiency Syndrome; nitazoxanide; Antiparasitic Agents
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; Diarrhea; Acquired Immunodeficiency Syndrome | interventions — nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide

SUMMARY:
The purpose of this study is to see if nitazoxanide (NTZ) can be used to treat AIDS patients suffering from cryptosporidiosis (diarrhea caused by the parasite Cryptosporidium).

DETAILED DESCRIPTION:
Patients receive oral nitazoxanide daily for 14 days, after which those with complete clinical and parasitologic response discontinue treatment. Non-responders and partial responders may continue therapy for an additional 14 days at the discretion of the physician. Non-responders who show signs of improvement or who have partial response after 28 days and those who relapse following complete response may continue therapy for an additional month, up to 60 days total. [AS PER AMENDMENT 10/30/96: Patients receive a daily treatment for 4 weeks, with subsequent dose escalation in the absence of drug-related toxicity. Patients who exhibit complete response after 2 months may continue at a maintenance dose. Patients enrolled after October 15, 1996 are randomized to 1 of 2 doses, with subsequent escalations made in the absence of toxicity. Complete responders may continue therapy at a maintenance dose and duration determined by the investigator. Non-responders after 6 months of therapy have treatment discontinued.] [AS PER AMENDMENT 8/5/97: All patients are evaluated at Weeks 1, 2, 4, and monthly thereafter.] [AS PER AMENDMENT 8/17/99: New patients start therapy on a different dosage of nitazoxanide. Those who do not respond after 4 weeks of therapy will escalate to a higher dosage. Patients who show a complete response at 2 consecutive visits (2 weeks apart) discontinue nitazoxanide therapy and go to follow-up.] [AS PER AMENDMENT 2/3/00: The Week 1 clinical evaluation is deleted from the study procedures.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 3 to 65 years old (need consent of parent or guardian if under 18).
* Have AIDS.
* Have a CD4 count less than or equal to 200 cells/mm3. (Note: Patients with a CD4 count greater than 200 cells/mm3 but who have had cryptosporidiosis for at least 4 weeks may be eligible for this study.)
* Test positive for the parasite Cryptosporidium and have severe diarrhea (at least 4 bowel movements per day) for at least 2 weeks.
* Have received treatment for cryptosporidiosis but have become reinfected after treatment.
* Agree to practice abstinence or use effective methods of birth control (such as a condom) before and during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant.
* Are infected with certain other parasites.
* Have a history of certain intestinal diseases.
* Have received certain medications.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Romark Laboratories LC, Tampa, Florida, United States